CLINICAL TRIAL: NCT05381857
Title: Genetic & Environmental Determinants Of Immune Phenotype Variance: A Longitudinal Assessment
Acronym: MI-V3
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-062
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy Subjects
Keywords: Immune response; Immune system; genotype-to-phenotype association; genetic variability; reference-based population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, urine, nasal swab, fecal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individual from the initial Milieu Intérieur study: Individual who provided samples for the initial Milieu Intérieur study
  Interventions: Other: Human Biological Samples

INTERVENTIONS:
Other: Human Biological Samples — Blood, urine, nasal swab, fecal samples

SUMMARY:
Effects of aging, genetics and environmental exposures on immune variation in a previously well-defined healthy population (NCT03905993).

DETAILED DESCRIPTION:
Susceptibility to infections, disease severity, and response to medical therapies and vaccines are highly variable from one individual to another.

Individual heterogeneity in the immune response can have an enormous impact on the likelihood to respond to therapy or the development of side effects secondary to vaccine administration. Because of the complexity of immune responses in the individual and within the population, it has not been possible thus far to define the parameters (genetic or environmental) that constitute a healthy immune system and its natural occurring variability.

The overall aim of the Milieu Intérieur study (NCT03905993) is to define the parameters that characterise a healthy immune response and its natural variation across individuals, and in doing so, inform clinical strategies for managing disease. To achieve this, in 2012, a total of 1000 healthy volunteers, descendants of mainland French persons for at least three generations, split equally by sex (1:1 sex ratio) and stratified across five-decades of life were recruited.

With the first data collection (clinical study), key fundamental insights were gained. The project has also established a rich sample and data repository, supporting ongoing integrative research in systems immunology and personalized medicine.

To provide a longitudinal assessment of the immune variation observed in the Milieu Intérieur cohort, this research aim to perform a follow-up study of the cohort, 10 years after the initial study.

ELIGIBILITY:
Inclusion Criteria:

* Any individual that provided samples for the initial Milieu Intérieur study (NCT03905993)
* Ability to give their informed consent in writing
* Subjects who, according to the investigator, can and will comply with the requirements of the protocol.
* Affiliated to the French social security or assimilated regimens

Exclusion Criteria:

* Individuals benefiting from a legal protection measure
* Individuals unable to express informed consent for participation
* Pregnant and breastfeeding women

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults subjects, aged from 30 to 79 years old that provided samples for the initial Milieu Intérieur study
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Identify associations with immune response variability | 20 years
  Identifying factors (genetic, epigenetic, immunological and environmental) that contributes to the observed heterogeneity in immune responses at the individual and population level over time

CONTACTS AND LOCATIONS:
Overall Officials: Lluis QUINTANA MURCI, PhD, Study Director — Institut Pasteur; Darragh DUFFY, PhD, Study Director — Institut Pasteur
Locations (1):
- Biotrial, Rennes, France

REFERENCES:
- [Background] Thomas S, Rouilly V, Patin E, Alanio C, Dubois A, Delval C, Marquier LG, Fauchoux N, Sayegrih S, Vray M, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. The Milieu Interieur study - an integrative approach for study of human immunological variance. Clin Immunol. 2015 Apr;157(2):277-93. doi: 10.1016/j.clim.2014.12.004. Epub 2015 Jan 3. PMID 25562703
- [Background] Duffy D, Rouilly V, Libri V, Hasan M, Beitz B, David M, Urrutia A, Bisiaux A, Labrie ST, Dubois A, Boneca IG, Delval C, Thomas S, Rogge L, Schmolz M, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Functional analysis via standardized whole-blood stimulation systems defines the boundaries of a healthy immune response to complex stimuli. Immunity. 2014 Mar 20;40(3):436-50. doi: 10.1016/j.immuni.2014.03.002. PMID 24656047
- [Background] Patin E, Hasan M, Bergstedt J, Rouilly V, Libri V, Urrutia A, Alanio C, Scepanovic P, Hammer C, Jonsson F, Beitz B, Quach H, Lim YW, Hunkapiller J, Zepeda M, Green C, Piasecka B, Leloup C, Rogge L, Huetz F, Peguillet I, Lantz O, Fontes M, Di Santo JP, Thomas S, Fellay J, Duffy D, Quintana-Murci L, Albert ML; Milieu Interieur Consortium. Natural variation in the parameters of innate immune cells is preferentially driven by genetic factors. Nat Immunol. 2018 Mar;19(3):302-314. doi: 10.1038/s41590-018-0049-7. Epub 2018 Feb 23. PMID 29476184
- See also: The website provides a description of the Milieu Intérieur project, consortium and collaborative studies — http://www.milieuinterieur.fr